CLINICAL TRIAL: NCT03928106
Title: Impact of Pharmacists Directed Medication Reconciliation on Reducing Medication Discrepancies in a Surgery Ward in an Educational Hospital in Jordan
Brief Title: Impact of Pharmacists Directed Medication Reconciliation on Reducing Medication Discrepancies in a Surgery Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Khawla Abu Hammour, Dr Associate professor (Principal Investigator), University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 65/2017
Record Dates: First submitted 2018-07-30; First posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Safety Issues
Keywords: Medication Reconciliation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Other): pharmacist responsible for enrollment will administer the following interventions: identifying the medication discrepancies make the recommendations to correct these discrepancies contact the physician to resolve these discrepancies
  Interventions: Other: pharmacists' recommendation
- control (Other): pharmacists will identify medication discrepancies no recommendation will be written by pharmacists to solve these discrepancies
  Interventions: Other: pharmacists' recommendation

INTERVENTIONS:
Other: pharmacists' recommendation — For patients in the intervention group, upon identification of drug discrepancies, pharmacist responsible for enrollment will be intervened by contacting the responsible clinician using a structured written consult form. The number of accepted recommendations by the clinicians will be documented and recorded. When the researcher suggests resolving an identified discrepancy and the responsible clinicians accept the suggestion will be called an accepted recommendation (just an acceptance without any correction), if the accepted suggestion is implemented then this will be called implemented recommendation.

SUMMARY:
Several previous studies have investigated the impact of a pharmacists-provided medication reconciliation service on medication discrepancies in the hospital settings Results showed that pharmacists were able to identify a range of 1.5-2.3 unintentional discrepancies per patient, leading to a significant reduction of 40-75% of the total identified medication discrepancies. No previous study has investigated the outcomes of involving the clinical pharmacist in a medication reconciliation service in in Jordan.

Acknowledging the importance of evaluating the value of medication reconciliation services in the different healthcare settings, this study is designed with the aim to evaluate the effect of pharmacists directed services (reconciliation plus counseling) on reducing medication discrepancies and improving patient's outcomes at discharge.

DETAILED DESCRIPTION:
Impact of Pharmacists Directed Medication Reconciliation on Reducing Medication Discrepancies in a Surgery Ward in an Educational Hospital in Jordan

1. Introduction Medication reconciliation is a technique used by healthcare providers at different care settings in order to prevent medication errors. According to the Institute for Safe Medication Practices Canada, medication reconciliation is defined as "a formal process in which healthcare providers work together with patients, families and care providers to ensure accurate and comprehensive medication information is communicated consistently across transitions of care". ISMP Canada has described the process of medication reconciliation as " a systematic and comprehensive review of patient's Best Possible Medication History (BPMH) to identify any possible medication discrepancies and to inform and enable prescribers to make the most appropriate prescribing decisions for the patient to solve identified discrepancies".

   Pharmacists are the healthcare providers responsible for providing optimal pharmaceutical care services. Regular medication review and medication reconciliation, beside the development of patient care plan, are considered as important pharmaceutical care tools.The Institute of Medicine reports acknowledged pharmacists as an essential resource of information on medication safe use, and their vital participation during hospital rounds as it improves medication safety.

   Currently, all hospitals have a pharmacy department to ensure that all patients receive their medications in the correct way by implementing the eight rights of medication administration (right patient, right medication, right dose, right route, right time, right documentation, right reason and right response). Clinical pharmacists can ideally influence physicians on their prescribing of medicines because they have the appropriate knowledge regarding therapeutics and are in continuous contact with them.Pharmacists have an important role in reducing discharge medical errors and patients' re-hospitalization.[6] Clinical pharmacists were found aware of the importance of their role in providing medication reconciliation.

   Several previous studies have investigated the impact of a pharmacists-provided medication reconciliation service on medication discrepancies in the hospital settings Results showed that pharmacists were able to identify a range of 1.5-2.3 unintentional discrepancies per patient, leading to a significant reduction of 40-75% of the total identified medication discrepancies. No previous study has investigated the outcomes of involving the clinical pharmacist in a medication reconciliation service in in Jordan.

   Acknowledging the importance of evaluating the value of medication reconciliation services in the different healthcare settings, this study is designed with the aim to evaluate the effect of pharmacists directed services (reconciliation plus counseling) on reducing medication discrepancies and improving patient's outcomes at discharge.
2. Methods 2.1. Study Design, participants and clinical setting This randomized controlled study will be conducted over three months at the Jordan University Hospital (JUH), a 550 beds tertiary teaching hospital located in Amman, the capital of Jordan.

Methods:

During the study period, 128 patients who fulfilled the inclusion criteria will be approached and asked to participate in the study. Inclusion criteria are: age ≥18 years; using at least 4 regular pre-admission medications; with more than 48 hours expected length of stay in the hospital; speaks Arabic; has no cognitive deficiency, and not involved in any other clinical trial. Patients will be excluded if they were in isolation; discharged within 24 hours of admission; discharged against medical advice; unable or unwilling to provide written informed consent; unable to provide a personal phone number; also patients who were enrolled were ineligible for re-inclusion in the study if they were admitted to JUH a second time during the study period.

Ethical approval from the Institutional Review Board (IRB) at the Jordan University Hospital (JUH) was obtained (Reference number: 65/2017).

2.2 Sample Size Calculation Setting alpha at 0.05, power of 80%, and using effect size of 0.5 (medium value), the minimum Required sample size to obtain a significant difference was calculated as 64 subjects per group.

Taking into account the possibility for dropout during the study period, a sample size of 128 patients is selected in this study.

2.3 Data collection and identification of medication discrepancies Patients will be recruited from all internal medicine department subdivisions at JUH. For each recruited patient, a pre-prepared validated data collection form will be used for data collection.Patients' specific data including demographic data, administrative data, medical related data, and BPMH. BPMH including pre-admission medications will be collected from the patients' medical records, followed by interviewing the patient (or their caregivers), and finally by interviewing the responsible clinicians (details about data collection are presented in a previously published study. For each patient, comorbidity will be calculated using Charlson Comorbidity Index (CCI). This index represents a tool that will be used to predict the ten year mortality rate in individuals with comorbid conditions.

Following data collection, a comparison between patients' current admission medications and patient's pre-admission medications will be done to identify any discrepancies between the two medication lists. Discrepancies will be categorized into dose discrepancies, frequency discrepancies, addition of a new drug, duplication of drugs, omission of drugs, or using wrong drugs.

Identified discrepancies will then be classified into documented or undocumented discrepancies. Documented discrepancies are defined as any change in medications that was justified in the patient's medical file. If the discrepancy is undocumented, the pharmacist will review the differences with the clinician in order to verify if the changes are intentional or made by error. In case of intentional discrepancies, the problem will be recorded as a 'documentation error'. Otherwise, unintentional discrepancies will be considered as 'medication errors'.

Unintentional discrepancies (medication errors) are classified into three classes based on the level of their seriousness as described by Cornish and others: "class 1 discrepancies are those unlikely to cause patient discomfort or clinical deterioration. Class 2 discrepancies are those with the potential to cause moderate discomfort or clinical deterioration, and class 3 discrepancies are those with the potential to cause severe discomfort or clinical deterioration". Discrepancies are classified by the two researchers of the study, and in the case of disagreement on classification, the discrepancy will be discussed until consensus is reached.

2.4 Pharmacist delivered intervention Following medication discrepancy identification, patients will be divided randomly into two groups, intervention and control. Patients will be assigned to their groups based on Statistical Package for Social Science (SPSS) version 22 generated random table for assignment (SPSS Inc., Chicago, IL, USA) (Figure 1).

For patients in the intervention group, upon identification of drug discrepancies, pharmacist responsible for enrollment will be intervened by contacting the responsible clinician using a structured written consult form. The number of accepted recommendations by the clinicians will be documented and recorded. When the researcher suggests resolving an identified discrepancy and the responsible clinicians accept the suggestion will be called an accepted recommendation (just an acceptance without any correction), if the accepted suggestion is implemented then this will be called implemented recommendation.

At discharge, the number of medication discrepancies will be assessed again for both groups. Also, the pharmacist provided intervention group patients with education about their medications, including: information about efficacy/side effects of medications, proper use and storage of medications, the importance of adherence, medication changes will be made while in hospital (i.e. reviewing pre-admission medications vs. medications at discharge).

The evaluation of carry-over effect of pharmacists' intervention on the number of discrepancies over months will be also assessed.

2.5 Statistical analysis Data will be entered and analyzed using Statistical Package for Social Science (SPSS) version 22 (SPSS Inc., Chicago, IL, USA). Descriptive analysis will be done using mean and standard deviation (SD) for continuous variables, and percentage for categorical variables. Checking for normality will be carried out using Shapiro-Wilk test, with P-value ≥ 0.05, indicating normally distributed continuous variables.

Group differences between control and intervention groups will be conducted using independent sample t-test/Mann Whitney U test (depending on data normality) or by using Chi-Square/Fisher exact test when appropriate. A paired t-test/Wilcoxon sign rank test will be performed to ascertain whether pharmacist's recommendations are effective in reducing the number of medication discrepancies An analysis of trend will be carried out using One-Way ANOVA to evaluate the trend in change of the number of discrepancies over the study period (to evaluate the carry-over study effect).

A P-value of less than 0.05 is considered statistically significant and all tests are two tailed.

6. Conflict of interest None of the authors have any conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* using at least 4 regular pre-admission medications
* more than 48 hours expected length of stay in the hospital
* speaks Arabic
* has no cognitive deficiency
* not involved in any other clinical trial

Exclusion Criteria:

* if they were in isolation
* discharged within 24 hours of admission
* discharged against medical advice
* unable or unwilling to provide written informed consent
* unable to provide a personal phone number
* patients who were enrolled were ineligible for re-inclusion in the study
* if they were admitted to JUH a second time during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
The number of accepted recommendations by the clinicians will be documented and recorded, an accepted recommendation, and implemented recommendation | From date of randomization until the date of first documented progression, assessed through study completion an average of 3 months
  The number of accepted recommendations by the clinicians will be documented and recorded, an accepted recommendation, implemented recommendation

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/22242793
- See also: Related Info — https://www.ismp-canada.org/medrec/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/15537552
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/17062324
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21763215
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/24327590
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/27198470
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/22471836
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/16585113
- See also: Related Info — http://erepository.uonbi.ac.ke/bitstream/handle/11295/98866/Okerosi_Prevalence%20And%20Risk%20Factors%20For%20Medication%20Discrepancies%20On%20Admission%20Of%20Elderly%20Diabetics%20At%20Kenyatta%20National%20Hospital,%20Kenya.pdf?sequence=1&isAllowed=y